CLINICAL TRIAL: NCT04437537
Title: A Pilot Study to Assess the Impact of PHOENIX Wound Matrix® on the Wound Microbiome in Chronic Diabetic Foot Ulcers
Brief Title: Pilot Study of PHOENIX Wound Matrix® Impact on Chronic DFU Wound Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenovoDerm (Industry)
Collaborators: Simon Tabchi DPM, PA Foot & Ankle Associates (Unknown); Lindsay Kalan PhD, Kalan Lab, McMaster University (Unknown)
Responsible Party: Sponsor
Organization: Nanofiber Solutions (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD2025-001.MB
Record Dates: First submitted 2020-05-23; First posted 2020-06-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer
Keywords: chronic diabetic foot ulcer; microbiome; PHOENIX Wound Matrix
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Phoenix Wound Matrix plus standard of care (Experimental): All subjects in this pilot study will receive Phoenix Wound Matrix in addition to the standard of care treatment for their diabetic foot ulcer.
  Interventions: Device: Bioresorbable 3D electrospun synthetic matrix

INTERVENTIONS:
Device: Bioresorbable 3D electrospun synthetic matrix — All participants in this study will receive PHOENIX Wound Matrix® in addition to the SOC treatment for their chronic DFU.
  Other Names: PHOENIX Wound Matrix®

SUMMARY:
A Pilot Study to Determine the Impact of the Phoenix Wound Matrix® on the Wound Microbiome in Chronic Diabetic Foot Ulcers

DETAILED DESCRIPTION:
The PHOENIX Wound Matrix® (PHOENIX) is a novel, fully synthetic and bioabsorbable advanced wound care device that provides a temporary microenvironment to support endogenous wound healing, allowing for the regeneration of functional, native tissue in the defect space/wound bed.

The human microbiome is a highly variable ecosystem comprising diverse microbiota of bacteria and fungi that vary more from one body site to another than from one individual to another, making it possible to define a "healthy microbiome core'' that occur frequently within different body sites. Perturbations of a body site's healthy microbiome core can disrupt the symbiotic relationship between host and associated microbes, resulting in pathogenicity and poor outcomes, such as chronic wounds.

The primary purpose of this study is to determine if PHOENIX alters the wound-associated microbiome in patients with chronic diabetic foot ulcers (DFUs).

Wound tissue and exudate samples in subjects with chronic DFUs will be collected and analyzed.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Subject is able and willing to provide consent, and Informed Consent Form is signed and dated prior to the initiation of any study-related activities.
2. 18 years of age or older.
3. Type 1 or type 2 diabetes mellitus.
4. At least one DFU that meet the following criteria:

   1. Ulcer is diagnosed as a partial- or full-thickness DFU located on the anatomical foot, defined as a minimum of 50% of ulcer area extending distal to the medial malleolus, excluding ulcers between the toes but including those of the heel.
   2. Wound surface area is ≥ 1 cm2 and ≤ 25 cm2 post-debridement at the time of Study Visit 1.
   3. Duration of the study ulcer will be a minimum of 4 weeks and no longer than 52 weeks at the time of the Study Visit 1.
   4. In the case of multiple ulcers, the largest ulcer meeting the study criteria will be designated the index ulcer and the only one included in the study. If other ulcerations are present on the same leg, there must be a margin of ≥ 2 cm between the index ulcer and all other ulcers, post-debridement.
   5. Wagner grade 1 or 2; or Wagner grade 3 with resolved abscess or osteomyelitis (confirmed by plain x-ray, bone biopsy, magnetic resonance imaging or bone scan) or resolved joint sepsis.
   6. Adequate vascular perfusion of the affected limb, confirmed by normal ankle pulses (posterior tibial and dorsalis pedis arteries). If pulse character is abnormal, ABI is required. Acceptable ABI results are ≤ 6 months old and must be within the specified range to qualify: 0.8 < ABI < 1.2.
5. Subject is willing and able to comply with offloading (as applicable for the location of the ulcer) or with use of appropriate footwear, as specified by the Investigator.
6. Subject is willing and able to comply with the requirements of this study, as instructed by the Investigator in accordance with the study protocol.

EXCLUSION CRITERIA:

1. Presence of signs and symptoms of infection at the index ulcer site or affected limb, including but not limited to cellulitis, osteomyelitis, excessive exudate, gangrene or deep tissue infection at the time of Study Visit 1.
2. Presence of diabetes with poor metabolic control as documented with an HbA1c ≥ 12.0 within 3 months of Study Visit 1.
3. Continued use of systemic antibiotics or use of systemic antibiotics within 7 days of Study Visit 1.
4. Females of childbearing potential.
5. Previous treatment with PHOENIX Wound Matrix®.
6. Participation in another clinical trial involving a device or systematically administered investigational study drug or treatment within 30 days of Study Visit 1 date.
7. Receiving or scheduled to receive a medication or treatment which, in the opinion of the Investigator, is known to interfere with, or affect, the rate and quality of wound healing.
8. History of bone cancer or metastatic disease of the affected limb, radiation therapy to the foot, or chemotherapy within the 12 months of Study Visit 1 date.
9. Treatment with wound dressings that include growth factors, engineered tissues, or skin substitutes within 30 days of Study Visit 1, or scheduled to receive such treatment during the Study.
10. Edema or lymphedema non-responsive to the standard of care.
11. Treatment with hyperbaric oxygen within 5 days of Study Visit 1 or scheduled to receive this treatment during the Study.
12. History of or intercurrent illnesses or conditions (other than diabetes) that would compromise the safety of the subject, or the normal wound healing process (i.e., end stage renal disease, immunosuppression, AIDS, bleeding disorders, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Wound Microbiome | From enrollment to the end of Study Visit 5 (4 weeks)
  Analysis of the wound microbiome in subjects with chronic DFUs prior to PHOENIX application and at follow-up Study Visits 3, and possibly 5 (if debridement is deemed necessary by the Investigator), again prior to the application of PHOENIX.
  This analysis will identify and quantify bacterial and fungal microorganisms present in the wound bed.

SECONDARY OUTCOMES:
Wound Biomarkers | From enrollment to the completion of Study Visit 5 (4 weeks)
  Wound fluid samples will be collected at Study Visits 1, 3, and possibly 5 (if debridement is required at Study Visit 5) for quantitative analysis of biomarkers of wound healing.
Wound Bed pH | From enrollment to completion of Study Visit 5 (4 weeks)
  Analysis of wound bed pH will be performed at all study visits upon removal of old dressings, prior to cleansing and debridement. During study visits where debridement is perform, pH will be analyzed post-debridement as well.

CONTACTS AND LOCATIONS:
Overall Officials: Simon G Tabchi, DPM, Principal Investigator — PA Foot & Ankle Associates; Lindsay Kalan, PhD, Principal Investigator — Kalan Lab, McMasters University; Elsa Englund Kayuha, MD, Study Director — RenovoDerm
Locations (1):
- PA Foot & Ankle Associates, Northampton, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study.

REFERENCES:
- [Background] A.G. Neto, R.A. Hickman, A. Khan, C. Nossa, Z. Pei, Chapter 1 - The Upper Gastrointestinal Tract-Esophagus and Stomach, Editor(s): Martin H. Floch, Yehuda Ringel, W. Allan Walker, The Microbiota in Gastrointestinal Pathophysiology, Academic Press, 2017, Pages 1-11, ISBN 9780128040249, https://doi.org/10.1016/B978-0-12-804024-9.00001-X.
- [Background] Kalan L, Grice EA. Fungi in the Wound Microbiome. Adv Wound Care (New Rochelle). 2018 Jul 1;7(7):247-255. doi: 10.1089/wound.2017.0756. PMID 29984114
- [Background] Grice EA, Kong HH, Conlan S, Deming CB, Davis J, Young AC; NISC Comparative Sequencing Program; Bouffard GG, Blakesley RW, Murray PR, Green ED, Turner ML, Segre JA. Topographical and temporal diversity of the human skin microbiome. Science. 2009 May 29;324(5931):1190-2. doi: 10.1126/science.1171700. PMID 19478181
- [Background] Ursell LK, Metcalf JL, Parfrey LW, Knight R. Defining the human microbiome. Nutr Rev. 2012 Aug;70 Suppl 1(Suppl 1):S38-44. doi: 10.1111/j.1753-4887.2012.00493.x. PMID 22861806
- [Background] Proctor LM. The Human Microbiome Project in 2011 and beyond. Cell Host Microbe. 2011 Oct 20;10(4):287-91. doi: 10.1016/j.chom.2011.10.001. PMID 22018227